CLINICAL TRIAL: NCT05744466
Title: A Real-world, Prospective, Observational Study of the Comparative Effectiveness of Deucravacitinib Versus Apremilast in Adults With Plaque Psoriasis - North American Region
Brief Title: A Real-world Observational Study to Compare Effectiveness of Deucravacitinib Vs Apremilast in Adults With Plaque Psoriasis
Acronym: RePhlect
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1105
Record Dates: First submitted 2023-01-30; First posted 2023-02-27 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Psoriasis
Keywords: Real-world; Deucravacitinib; Observational
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib; apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants that have initiated deucravacitinib
  Interventions: Drug: Deucravacitinib
- Cohort 2: Participants that have initiated apremilast
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Deucravacitinib — As prescribed by treating clinician
  Groups: Cohort 1
Drug: Apremilast — As prescribed by treating clinician
  Groups: Cohort 2

SUMMARY:
The purpose of this study is to understand the comparative effectiveness of deucravacitinib versus apremilast in adults with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with plaque psoriasis by a dermatologist
* Newly initiating an eligible medication for enrollment (i.e., deucravacitinib, apremilast)
* Actively enrolled in the CorEvitas Psoriasis Registry and have documented consent to allow copies of information from the registry be used for research purposes

Exclusion Criteria:

* Participation (current or planned) in an interventional clinical trial (does not include observational registry or study)
* Restart of treatments with the study eligible therapies previously received at any time during the participants' treatment history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with moderate-to-severe plaque psoriasis who initiate deucravacitinib or apremilast within the CorEvitas Psoriasis Registry will be enrolled. Participants will be followed every 6 months from initiation up to 5 years or discontinuation, whichever occurs first. This is a real-world study and hence the follow-up are done based on the clinical practice done by dermatologists.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in body surface area (BSA) | At baseline and every 6 months up to 60 months or treatment discontinuation
Investigator global assessment (IGA) response 0/1 | Up to 60 months
Dermatology life quality index (DLQI) response 0/1 | Up to 60 months
Time from date of treatment initiation to date of discontinuation | Up to 60 months

SECONDARY OUTCOMES:
75 percent improvement in Psoriasis area and severity index (PASI) score | At baseline and every 6 months up to 60 months or treatment discontinuation
PASI score response ≤ 3 | At baseline to follow-up, up to 60 months
PASI score response ≤ 5 | At baseline to follow-up, up to 60 months
PASI score change from baseline | At baseline to follow-up, up to 60 months
National psoriasis foundation (NPF) acceptable body surface area (BSA) response | At baseline to follow-up, up to 60 months
NPF target BSA response | At baseline to follow-up, up to 60 months
BSA ≤3% | At baseline to follow-up, up to 60 months
Change in investigator global assessment (IGA) score | Up to 60 months
Change in dermatology life quality index (DLQI) response | At baseline to follow-up, up to 60 months
Change in DLQI response ≤5 | At baseline to follow-up, up to 60 months
Change in visual analog scale (VAS): Itch response | At baseline to follow-up, up to 60 months
Change in VAS: Skin Pain response | At baseline to follow-up, up to 60 months
Change in VAS: Fatigue Response | At baseline to follow-up, up to 60 months
Merit-based Incentive Payment System (MIPS) Clinical Response to Oral Systemic or Biologic Medications | At baseline to follow-up, up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts